CLINICAL TRIAL: NCT06504459
Title: A Phase II Study of Venetoclax (ABT-199) in Combination With Cladribine and Low-Dose Cytarabine Alternating With Azacitidine Plus Venetoclax in Newly Diagnosed Monocytic AML and Active-Signaling Mutated AML
Brief Title: Venetoclax in Combination With Cladribine and Cytarabine Alternating With Azacitidine Plus Venetoclax for the Treatment of Newly Diagnosed Monocytic AML and Active Signaling Mutated AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); AbbVie (Industry)
Responsible Party: Principal Investigator, Curtis Lachowiez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00026216; NCI-2024-05084 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00026216 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-07-11; First posted 2024-07-16 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Acute Monocytic Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute | interventions — Azacitidine; Specimen Handling; Biopsy; Cladribine; Cytarabine; Spinal Puncture; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, cladribine, cytarabine, azacitidine) (Experimental): See Detailed Description
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cladribine; Drug: Cytarabine; Procedure: Echocardiography; Procedure: Lumbar Puncture; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; Spinal Tap
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Other: Questionnaire Administration — Ancillary studies
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial tests how well venetoclax with cladribine and cytarabine alternating with azacitidine and venetoclax works in treating patients with newly diagnosed monocytic acute myeloid leukemia (AML) and active signaling mutated AML. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking BCL-2, a protein needed for cancer cell survival. Chemotherapy drugs, such as cladribine, cytarabine and azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax with cladribine and cytarabine alternating with azacitidine and venetoclax may kill more cancer cells in patients with newly diagnosed monocytic AML and active signaling mutated AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess efficacy of the investigational treatment based on disease remission.

SECONDARY OBJECTIVES:

I. Assess efficacy of the investigational treatment based on clinical response. II. Assess any-cause survival after treatment. III. Assess survival in the absence of treatment failure, hematologic relapse, or progressive disease.

IV. Assess duration of response, based on morphological assessments. V. Assess the safety and tolerability of the regimen.

EXPLORATORY OBJECTIVES:

I. Assess response based on measurable residual disease (MRD). II. Identify markers of clonal or clinical response and resistance to treatment.

III. Assess participant quality of life (QoL) using Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO CTCAE).

OUTLINE:

INDUCTION: Patients receive cladribine intravenously (IV) over 1-2 hours on days 1-5, cytarabine subcutaneously (SC) twice daily (BID) on days 1-10, and venetoclax orally (PO) once daily (QD) on days 1-21 of cycle 1.

RE-INDUCTION: Patients with > 5% blasts after cycle 1 receive cladribine IV over 1-2 hours on days 1-5, cytarabine SC BID on days 1-10, and venetoclax PO QD on days 1-21 of cycle 2.

REMISSION AFTER INDUCTION: Patients who achieve complete remission (CR)/CR with partial hematologic recovery/CR with incomplete blood count recovery/morphologic leukemia-free state (MLFS) after cycle 1 of induction, receive cladribine IV over 1-2 hours on days 1-3, cytarabine SC BID on days 1-10 and venetoclax PO QD on days 1-21 of cycle 2.

CONTINUING THERAPY: Patients who achieve MLFS receive venetoclax PO QD on days 1-21 and azacitidine IV or SC QD on days 1-7 for 2 cycles then cladribine IV over 1-2 hours on days 1-3, cytarabine SQ BID on days 1-10 and venetoclax PO QD on days 1-21 for 2 cycles. Cycles repeat every 28 days and continue to alternate every 2 cycles for up to cycle 18 in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) as clinically indicated on study. Patients also undergo bone marrow aspiration and biopsy and blood sample collection throughout the study.

At completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend the investigational nature of the study and provide informed consent (i.e., participant or legally authorized representative [LAR]). Written informed consent must be obtained prior to any study-specific procedures or interventions

  • Sign informed consent for the #4422 Biorepository prior to any study-specific procedures of interventions
* Eligible AML patients of all races and ethnic groups will be considered for participation, irrespective of gender identity
* Newly diagnosed, histologically confirmed monocytic AML, as defined by World Health Organization (WHO), or active signaling mutated AML defined as AML with mutation(s) to N/KRAS, FLT3 ITD/TKD, NF1, PTPN11 or CBL
* Ineligible for standard of care induction therapy using intensive chemotherapy (IC) or unwilling to undergo IC induction therapy. Ineligible for IC is defined as

  * ≥ 75 yrs of age; OR
  * 18-74 yrs of age with one of the following:

    * Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 2 at screening
    * Severe cardiac disorder (e.g., congestive heart failure requiring treatment, ejection fraction ≤ 50%, or chronic stable angina)
    * Severe pulmonary disorder (e.g., diffuse capacity of the lung for carbon monoxide [DLCO] ≤ 65% or forced expiratory volume in 1 second [FEV1] ≤ 65%)
    * Creatinine clearance < 45 ml/min (calculated by the Cockcroft-Gault equation)
    * Hepatic disorder with total bilirubin > 1.5 x upper limit of normal (ULN)
    * Any other comorbidity that the treating physician judges to be incompatible with IC
* If ≥ 75 yrs of age, the following organ function values must be met and ECOG must be 0 to 2 at screening:

  * Creatinine clearance (calculated with the Cockcroft-Gault equation) ≥ 30 ml/min
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (Unless due to leukemic infiltration)
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x ULN (Unless due to leukemic infiltration) (With the exception of documented Gilbert's syndrome or similar conditions. Liver function testing (LFT) and timepoints may be added, as clinically indicated, in such cases)

    * Note: In cases of confirmed leukemic organ involvement, exceptions may be made
* Willing and able to provide bone marrow (BM) samples, including BM samples for research use only analysis
* Willing and able to accept supportive and prophylactic care for hematologic toxicities, infection, and immediate sequalae
* Willingness to adhere to (a) study schedule of activities; (b) requirements for bio samples collections; and (b) lifestyle restrictions while on-treatment
* Negative urine pregnancy test at screening and within 24 hours of cycle 1 day 1 (C1D1) for persons of childbearing potential (PCBP). Serum pregnancy testing will be used for confirmation in cases of equivocal results. Pregnancy is exclusionary because the agents used in this study have the potential for teratogenic or abortifacient effects
* Willingness to comply with study requirements for contraception within the specified timeframe, as follows:

  * Sperm producing participants who are active with PCBP must use approved contraception from C1D1 to 30 days, 3 months, or 6 months, after the last dose of venetoclax (30 days), azacitidine (3 months), cladribine (6 months), or cytarabine (6 months), whichever is later in time
  * PCBP who are sexually active with sperm-producing persons must use contraception from C1D1 to 30 days after the last dose of venetoclax or to 6 months after the last dose of azacitidine, cladribine, or cytarabine, whichever is later in time

Exclusion Criteria:

* Symptomatic central nervous system involvement with AML
* Prior treatment for AML, with the exception of cytoreduction for proliferative disease (per institutional protocol) with any of the following: Hydroxyurea, hematopoietic growth factors, leukapheresis
* Another active malignancy within the previous 5 years of C1D1
* Investigational therapy within 28 days of C1D1, or within 5 half-lives or longer, if known
* Recent and significant medical interventions, such as major surgery within 28 days or stem cell transplant within 100 days (and without active treatment for graft versus host disease [GVHD]) of C1D1. Standard of care procedures for patients with hematologic malignancies, such as biopsies and lumbar punctures, are not exclusionary
* Hypersensitivity to any of the components of the investigational regimen (i.e., cladribine, cytarabine, venetoclax, azacitidine) or any excipients in the formulations
* Treatment based on agents targeting or inhibiting BCL-2 (for other, prior indication/malignancy) within the previous 5 years
* History of dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Use of drugs with documented drug-drug interaction toxicities with the study drugs

  * Strong or moderate CYP3A4 inducers or inhibitors within 2 days or 3 half lives whichever is longer, prior to C1D1 are exclusionary. Dose adjustments and other modifications may be considered if the wash-out period has not been met, with the approval of the investigator and the research pharmacy
* Uncontrolled infection. Participants with controlled infection must be afebrile and hemodynamically stable for at least 72 hours prior to C1D1 and must be amenable to alternate treatment if current treatment will interact with investigational regimen
* Active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV). Enrollment of individuals with evidence of chronic HBV or HCV infection will be considered on a case-by-case basis by the principal investigator
* Individuals with serology positive for human immunodeficiency virus (HIV) and under active treatment with highly active antiretroviral therapy (HAART) (or another therapy that may interfere with metabolism of study agents)
* Pregnancy at enrollment or unwillingness to stop breastfeeding. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding be discontinued from start of treatment until 1 week after the final dose of any study drug
* Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, unstable cardiac or pulmonary function or acute insufficiency (e.g., symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia), or psychiatric illness or social situation that could limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2027-10-11 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission (CRc) rate | At start of treatment to post-induction disease assessment (Cycle 1 Day 21 or Cycle 2 Day 21. Each cycle is 28 days)
  CRc is defined as achievement of complete remission (CR), CR with partial hematologic recovery (CRh) or CR with incomplete blood count recovery (CRi) after induction (or re-induction). The CRc rate will be computed on the safety set and presented with a point-estimate and exact binomial 95% confidence interval (CI). CRc will also be modeled with univariable logistic regressions, applied to the efficacy set, to determine if any baseline patient or disease feature is correlated with clinical response.

SECONDARY OUTCOMES:
Overall response rate (ORR) | At start of treatment to post-induction disease assessment (Cycle 1 Day 21 or Cycle 2 Day 21. Each cycle is 28 days)
  ORR will be defined as the proportion of evaluable participants who attain a partial remission (PR) or better (i.e., CR, CRh, CRi, morphologic leukemia-free state [MLFS], or PR) while on investigational treatment. ORR will be computed for both the safety set and the efficacy set and presented with a point estimate and exact binomial CI. ORR will also be modeled with univariable logistic regressions with baseline patient and disease features as predictors and results considered hypothesis-generating.
Overall survival (OS) | At start of treatment to death up to 2 years
  OS will be computed for both the safety set and the efficacy set, and estimated with the Kaplan-Meier method. Median OS and OS rates at common landmark times (e.g., 1 year, 2 years) will be estimated with 95% log-log CIs. For both sets, univariable Cox models will be fit to OS to assess the impact of baseline patient and disease features with results (i.e., unadjusted hazard ratios and Wald test p-values) considered hypothesis-generating. Median follow-up will utilize a patient's OS measurement and censoring status and be estimated using the reverse Kaplan-Meier method.
Event-free survival (EFS) | At start of treatment to primary refractory disease, hematologic relapse, discontinuation of treatment due to toxicity, disease progression or death up to 2 years
  EFS will be measured from start of treatment to the earliest date of treatment failure, progressive disease, or death from any cause. EFS will be estimated for the efficacy set using the Kaplan-Meier method, with median EFS and EFS rates at common landmark times presented with 05% log-log CIs. EFS will be alternatively estimated upon assigning 1-day event times to participants who never achieve MLFS or better. Univariable Cox models will be fit to EFS to assess the impact of baseline patient and disease features with model results considered hypothesis-generating.
Duration of response (DOR) | At first date of documented ≥ MLFS or better to primary refractory disease, hematologic relapse, discontinuation of treatment due to toxicity, disease progression or death up to 2 years
  DOR will be measured from the first date of documented hematologic response to the earliest of the following occurrences: hematologic relapse, disease progression (clinical or morphologic), or any-cause death. DOR will be estimated by the Kaplan-Meier method. Median DOR will be presented with a 95% log-log CI.
Incidence of grade ≥ 3 adverse events (AEs) | At start of treatment up to 30 days after last dose of any study drug
  AEs severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Percentage of patients achieving 80% relative dose intensity | At start of treatment to end of treatment up to 1 year and 5 months
  The percentage of participants achieving 80% relative dose intensity will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Curtis A Lachowiez, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States